CLINICAL TRIAL: NCT01754480
Title: A Prospective, Single-blind, Randomized, Phase III Study to Evaluate the Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) as an Adjunct to Hemostasis During Parenchymous Tissue Open Surgeries
Brief Title: Safety and Efficacy of Fibrin Sealant Grifols (FS Grifols) During Parenchymous Tissue Open Surgeries
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Biologicals, LLC (Industry)
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: IG1102
Record Dates: First submitted 2012-12-18; First posted 2012-12-21 (Estimated); Results first posted 2017-02-08 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Parenchymous Tissue Surgical Bleeding
Keywords: Fibrin Sealant; Parenchymous tissue open surgery; Hepatic Resection; Oxidized cellulose pads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fibrin Sealant Grifols (Experimental): Fibrin Sealant Grifols consisting of 3 mL fibrinogen and 3 mL thrombin in separate syringes assembled on a syringe holder (6 mL of solution in total).
  Interventions: Biological: Fibrin Sealant Grifols
- Surgicel® (Active Comparator): Surgicel® is a sterile, absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose.
  Interventions: Device: Surgicel®

INTERVENTIONS:
Biological: Fibrin Sealant Grifols — Combination of 3 mL fibrinogen and 3 mL thrombin, in separate syringes assembled on a syringe holder (6 mL of solution in total), applied topically to the target bleeding site.
  Arms: Fibrin Sealant Grifols
Device: Surgicel® — Up to four Surgicel® sheets applied to the target bleeding site according to Package Insert instructions and the surgeon's usual clinical practice.
  Other Names: Fibrillar absorbable hemostat; Oxidized regenerated cellulose hemostat
  Arms: Surgicel®

SUMMARY:
This study is designed to assess the safety and efficacy of Fibrin Sealant Grifols in patients undergoing open surgical procedures where bleeding may be present on parenchymous tissue (e.g., solid abdominal organs such as the liver). The purpose of this study is to demonstrate that Fibrin Sealant Grifols is not inferior to commercially-available oxidized cellulose pads (Surgicel®) in providing benefit in the time to hemostasis (i.e, the stoppage of bleeding). This study has a Preliminary Part (I) for study teams to become familiar with the application of Fibrin Sealant Grifols and to assess safety and a Primary Part (II) to assess the safety and efficacy of Fibrin Sealant Grifols. In both parts of the study, patients will be randomized in a 1:1 ratio to either Fibrin Sealant Grifols or Surgicel.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin (Hgb) ≥ 8.0 g/dL at Baseline (within 24 hours prior to surgical procedure).
* Require elective (non-emergency), open (non-laparoscopic), hepatic resection (anatomic or non-anatomic resections of at least one anatomical hepatic segment, or equivalent tissue volume).
* A target bleeding site can be identified.
* Target bleeding site is identified on the cut raw liver surface (resection area).
* Target bleeding site has moderate bleeding according to the Investigator's judgment.

Exclusion Criteria:

* Require hepatic resection due to trauma.
* Infection in the anatomic surgical area.
* History of severe (e.g. anaphylactic) reactions to blood or to any blood-derived product.
* Previous known sensitivity to any Fibrin Sealant Grifols component or any Surgicel® component.
* Females who are pregnant or nursing a child at Baseline (within 24 hours prior to surgical procedure).
* Receiving an organ transplant during the same surgical procedure.
* Undergone a therapeutic surgical procedure within 30 days from the screening visit.
* A target bleeding site cannot be identified.
* The target bleeding site has a mild or severe bleeding.
* Occurrence of major intraoperative complications that require resuscitation or deviation from the planned surgical procedure.
* Application of any topical haemostatic material on the resection surface of the liver prior to application of study treatment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (33):
- United States (26):
  - 224, Loma Linda, California
  - 214, Los Angeles, California
  - 213, New Haven, Connecticut
  - 223, Augusta, Georgia
  - 228, Chicago, Illinois
  - 227, Goshen, Indiana
  - 207, Louisville, Kentucky
  - 220, New Orleans, Louisiana
  - 229, Bethesda, Maryland
  - 201, St Louis, Missouri
  - 231, Las Vegas, Nevada
  - 200, Albany, New York
  - 211, New York, New York
  - 212, New York, New York
  - 230, Charlotte, North Carolina
  - 233, Cincinnati, Ohio
  - 400, Hershey, Pennsylvania
  - 218, Philadelphia, Pennsylvania
  - 204, Philadelphia, Pennsylvania
  - 205, Charleston, South Carolina
  - 217, Memphis, Tennessee
  - 206, Nashville, Tennessee
  - 216, 219, Houston, Texas
  - 232, Salt Lake City, Utah
  - 226, Charlottesville, Virginia
  - 202, Madison, Wisconsin
- Hungary (2):
  - 602, Budapest
  - 600, Pécs
- Russia (2):
  - 640, Moscow
  - 641, Saint Petersburg
- Serbia (3):
  - 621, 622, 623, Belgrade
  - 620, 625, Niš
  - 624, Novi Sad

RESULTS

PARTICIPANT FLOW:
Groups:
- Surgicel®: Surgicel® is a sterile, absorbable knitted fabric prepared by the controlled oxidation of regenerated cellulose. Up to four Surgicel® sheets applied to the target bleeding site according to Package Insert instructions and the surgeon's usual clinical practice.
Period: Part I + Part II (Overall Study)
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Started | 163 | 162
Completed Study up to Week 6 | 147 | 153
Completed | 138 (Completed Virology follow-up visit at Month 3 or Month 6 (not required for 2 pediatric subjects)) | 139 (Completed Virology follow-up visit at Month 3 or Month 6 (not required for 3 pediatric subjects))
Not Completed | 25 | 23
Period: Primary Part II
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Started | 111 | 113
Completed Study up to Week 6 | 100 | 108
Completed | 96 (Completed Virology follow-up visit at Month 3 or Month 6 (not required for pediatric subjects)) | 102 (Completed Virology follow-up visit at Month 3 or Month 6 (not required for pediatric subjects))
Not Completed | 15 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fibrin Sealant Grifols | Surgicel® | Total
Number analyzed (Participants) | 163 | 162 | 325
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.82 (13.753) | 57.04 (15.194) | 57.93 (14.494)
Age, Customized [Number; unit: participants]
  <=11 years | 2 | 1 | 3
  Between 12 and 17 years | 0 | 2 | 2
  Between 18 and 64 years | 100 | 101 | 201
  >=65 years | 61 | 58 | 119
Gender [Count of Participants; unit: Participants]
  Female | 78 | 77 | 155
  Male | 85 | 85 | 170
Region of Enrollment [Number; unit: participants]
  Russian Federation | 3 | 2 | 5
  Hungary | 19 | 19 | 38
  United States | 88 | 91 | 179
  Serbia | 53 | 50 | 103

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Hemostasis by Four Minutes After Treatment Start
Description: Subjects achieving hemostasis at the target bleeding site by 4 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure.
Time Frame: From start of treatment until 4 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: Percent of subjects achieving hemostasis
Groups:
- Fibrin Sealant Grifols: Fibrin Sealant Fibrin Sealant Grifols: Combination of 3 mL fibrinogen and 3 mL thrombin, in separate syringes assembled on a syringe holder (6 mL of solution in total), applied topically to the target bleeding site.
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Number analyzed (Participants) | 111 | 113
Percent of subjects achieving hemostasis | 92.8 | 80.5

2. Secondary Outcome: Proportion of Subjects Achieving Hemostasis by Three Minutes After Treatment Start
Description: Subjects achieving hemostasis at the target bleeding site by 3 minutes following the start of treatment without the occurrence of re-bleeding until the completion of surgical closure.
Time Frame: From start of treatment until 3 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: Percent of subjects achieving hemostasis
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Number analyzed (Participants) | 111 | 113
Percent of subjects achieving hemostasis | 85.6 | 62.8

3. Secondary Outcome: Time to Hemostasis
Description: Time in minutes for achievement of hemostasis at the target bleeding site measured from the start of treatment until 10 minutes after treatment start.
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Number analyzed (Participants) | 111 | 113
minutes | 2.0 [2.00 to 3.00] | 3.0 [2.00 to 3.00]

4. Secondary Outcome: Cumulative Proportion of Subjects Having Achieved Hemostasis at the Target Bleeding Site by Specified Time Points
Description: Cumulative proportion of subjects having achieved hemostasis by each of the following time points:
  * At 2 minutes following start of study treatment
  * At 5 minutes following start of study treatment
  * At 7 minutes following start of study treatment
  * At 10 minutes following start of study treatment
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: Percent of subjects achieving hemostasis
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Number analyzed (Participants) | 111 | 113
Percent of subjects achieving hemostasis
  Hemostasis by 2 minutes | 55.9 | 41.6
  Hemostasis by 5 minutes | 97.3 | 85.0
  Hemostasis by 7 minutes | 97.3 | 87.6
  Hemostasis by 10 minutes | 98.2 | 92.0

5. Secondary Outcome: Prevalence of Treatment Failures
Description: Protocol-defined bleeding at the target bleeding site after the start of treatment or the use of alternative hemostatic treatments (with exception of reversal of heparin) or maneuvers at the target bleeding site after the start of treatment.
Time Frame: From start of treatment until 10 minutes after treatment start
Population: Efficacy analysis was performed on subjects in the Primary Part (II) of the study
Measure: Number; unit: percent of subjects
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Number analyzed (Participants) | 111 | 113
percent of subjects | 7.2 | 19.5

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the time informed consent was obtained through the Post-Operative Week 6 (±4 days) Visit
Arm/Group | Fibrin Sealant Grifols | Surgicel®
Serious Adverse Events (participants affected / at risk) | 30/163 | 23/162
Other Adverse Events (participants affected / at risk) | 131/163 | 136/162
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=163) | Surgicel® (N=162)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 2
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 2 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 2 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Device occlusion (General disorders) | 1 | 0
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 1
Biloma (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 1
Hepatic necrosis (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Portal vein thrombosis (Hepatobiliary disorders) | 1 | 0
Abdominal abscess (Infections and infestations) | 1 | 2
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Enterovirus infection (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Wound infection (Infections and infestations) | 1 | 0
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Post procedural bile leak (Injury, poisoning and procedural complications) | 4 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Venous injury (Injury, poisoning and procedural complications) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 1 | 0
Electrocardiogram ST segment abnormal (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain injury (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acute (Renal and urinary disorders) | 3 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Lung operation (Surgical and medical procedures) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 3 | 1
Embolism (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 1
Shock (Vascular disorders) | 1 | 0
Vena cava thrombosis (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fibrin Sealant Grifols (N=163) | Surgicel® (N=162)
Anaemia (Blood and lymphatic system disorders) | 21 | 26
Tachycardia (Cardiac disorders) | 14 | 24
Abdominal pain (Gastrointestinal disorders) | 10 | 3
Constipation (Gastrointestinal disorders) | 20 | 23
Nausea (Gastrointestinal disorders) | 34 | 38
Vomiting (Gastrointestinal disorders) | 13 | 17
Oedema peripheral (General disorders) | 14 | 11
Pyrexia (General disorders) | 16 | 19
Incision site pain (Injury, poisoning and procedural complications) | 12 | 11
Procedural haemorrhage (Injury, poisoning and procedural complications) | 9 | 4
Procedural pain (Injury, poisoning and procedural complications) | 59 | 61
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 11
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 15
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 11 | 10
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 11
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 12
Hypertension (Vascular disorders) | 14 | 12
Hypotension (Vascular disorders) | 21 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.